CLINICAL TRIAL: NCT00276120
Title: Identification of Novel Genetic Risk Factors That Contribute to the Risk for Breast Cancer
Brief Title: Identification of Novel Genetic Factors That Contribute to Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Amanda Toland, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-12164
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Invasive Breast Cancer
Keywords: Breast; Cancer; Young; Women
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify novel genetic factors which distinguish breast cancer in younger women compared to older women. By identifying these novel genetic factors we believe more specific therapies can be developed and breast cancer may be prevented among women with an increased cancer risk. A woman does not have to live in St. Louis to participate.

DETAILED DESCRIPTION:
Breast cancer takes its greatest toll on younger women, as it is the leading category of cancer deaths for women 20-39 years of age. Sadly, survival rates are lowest among women diagnosed at a young age. This impact is most significant among African-American women who have the highest incidence and mortality rate among women less than 45 years of age. The goal of our program is to identify the genetic factors which distinguish breast cancer in younger women compared to older women.

Women who were diagnosed with invasive breast cancer 40 years of age or younger are invited to participate. The age at diagnosis is used to determine eligibility, not a woman's current age. Women who have undergone genetic testing of the BRCA1, BRCA2, p53, pTEN, e-cadherin, or LKB1 genes are eligible to participate. Young women with breast cancer are asked to: sign a consent form, submit a sample of blood, release their cancer related records, and answer some family history questions.

We will use a family based case control approach in our analysis. As such, if a woman's parents are living, they will be invited to participate as a "comparison" group. The parents are asked to: sign a consent form, submit a sample of blood, and release any cancer records.

A woman does not have to live in St. Louis to participate. All study related materials can be mailed directly to the young woman or her parents. There is no expense to the family. All materials are kept strictly confidential and participation is completely voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with invasive breast cancer 40 years of age or younger. If their parents are living, the parents are also invited to participate, regardless of their history of cancer.

Exclusion Criteria:

* Women diagnosed with in-situ breast cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women diagnosed with invasive breast cancer < 40 years of age
Sampling Method: Probability Sample
Enrollment: 4385 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Toland, PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu